CLINICAL TRIAL: NCT05928546
Title: Efficacy of Quercetin Nanoemulgel as Adjunct Local Delivery Drug in Non-surgical Treatment of Periodontitis
Brief Title: Effect of Quercetin in Treatment of Periodontitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Alghriany, Lecturer, Oral medicine, Periodontology and Oral diagnosis, Faculty of dentistry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Quercetin in periodontitis
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Inflammation Gum
Keywords: Periodontitis; inflammation; Quarcetin; Nanoemulgel
MeSH Terms: conditions — Gingivitis; Periodontitis; Inflammation | interventions — Quercetin; Weights and Measures; Root Planing

STUDY DESIGN:
Intervention Model Description: Group(I): 10 sites will receive non-surgical periodontal therapy (scaling and root planing) . Group(Ⅱ): 10 sites will receive non-surgical periodontal therapy followed by the application of quercetin nanoemulgel local delivery 2 times one at the day of non-surgical periodontal therapy and after 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group(I):scaling and root planing only (Placebo Comparator): 10 sites will receive non-surgical periodontal therapy (scaling and root planing) .
  Interventions: Device: scaling and root planing
- Group(Ⅱ):scaling and root planing with application of quercetin nanoemulgel (Active Comparator): 10 sites will receive non-surgical periodontal therapy followed by the application of quercetin nanoemulgel local delivery 2 times one at the day of non-surgical periodontal therapy and after 2 weeks.
  Interventions: Drug: Quercetin; Device: scaling and root planing

INTERVENTIONS:
Drug: Quercetin — Intra-pocket application of quercetin nanoemulgel :
  * After conventional periodontal treatment, the teeth were isolated by cotton rolls for intra pocket application of the gel.
  * That gel was injected in periodontal pocket using syringe with blunt cannula till the gel excess exit from the pocket .
  Arms: Group(Ⅱ):scaling and root planing with application of quercetin nanoemulgel
Device: scaling and root planing — - Full-mouth scaling and root planing was performed in 1-2 sessions within 2 weeks using manual scalers and curettes or ultrasonic scaler and local anesthesia was used in case of need for patient comfort.

SUMMARY:
Periodontitis is an immune-inflammatory disease affecting the supporting structures of the teeth. It is a disease of multifactorial etiology, with microbial, genetic, environmental and host factors involved, with the release of oxygen-free radicals by the inflammatory cells. Quercetin, have shown potential antimicrobial activity, lowering of inflammatory markers, cholesterol reduction and inhibiting bone loss. However, this data has largely been obtained from in vitro and animal studies, but data from human studies are limited.

DETAILED DESCRIPTION:
Quercetin has been found to decrease the extracellular matrix degradation, promote wound healing when tested in gingival fibroblasts, and showed excellent antibacterial properties. It also possesses antioxidant effect which can be explored to restrict the inflammation in periodontitis. Despite the beneficial effects of Quercetin, its poor aqueous solubility and poor bioavailability result in limited absorption, so scientists have worked on improving the bioavailability of Quercetin using various approaches, such as nanosuspension , self-nano emulsifying systems , microemulsion , solid lipid nanoparticles and cyclodextrin complexes. The combination of oils and emulsifiers enhances the absorption of Quercetin. Hence, nanoemulsion could be a suitable drug delivery vehicle for the loading of Quercetin. Nanoemulsions are more beneficial than microemulsions, as they have high kinetic stability and a smaller droplet size. Therefore, the present study will investigate the efficacy of nanoemulgel of quercetin as adjunct to conventional therapy in treatment of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Patients with periodontitis stage ( Ⅰ & Ⅱ ). Stage I have CAL 1 to 2mm with no tooth loss and probing depth ≤4 mm. Stage II have CAL 3 to 4mm with no tooth loss and probing depth ≤5 mm..
  * Patients who have teeth with both mesial and distal neighboring teeth .
  * Patient with more than 20 natural teeth .
  * Patient free from any systemic disease that may effect the periodontal status according to the criteria of Cornell Medical Index and its modification.

Exclusion Criteria:

* Long-term therapy with medications within a month prior to enrollment that could affect periodontal status or healing.
* Pregnant woman and lactating mothers .
* Patients with a history of traumatic occlusion.
* Teeth with both endo-perio lesion .
* Patients with previous periodontal treatment including scaling and root planing and periodontal surgery in the last 3 and 6 months, respectively .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the changes in the clinical attachment loss | at base line, 1 month and 3 months after treatment
  Attachment level was measured using UNC15(University of North Carolina) periodontal probe. Clinical attachment loss was measured as the distance from the cemento-enamel junction to the base of the pocket.
Probing depth | at base line, 1 month and 3 months after treatment
  The measurement were recorded by UNC15(University of North Carolina) periodontal probe . Pocket depth was measured as the distances from the free gingival margin to the base of the periodontal pocket.
interferon IFN-γ analysis | at base line, 1 month and 3 months after treatment
  The samples were assayed for (IFN-γ) levels using commercially available enzyme-linked immune-sorbent assay (ELISA) . Highly sensitive ELISA kit was used to detect the (IFN-γ) level in pg/ml in the sample of GCF according to the manufacturer's instructions.
reactive oxygen species (ROS) | at base line, 1 month and 3 months after treatment
  The samples were assayed for antioxidant effect of quercetin using commercially available reactive oxygen species( ROS) kit . Highly sensitive ROS kit was used according to the manufacturer's instruction

SECONDARY OUTCOMES:
Plaque index (PI) | at base line, 1 month and 3 months after treatment
  It used to assess plaque accumulation around gingival margin.
  The degree of plaque accumulation was recorded as follow:
  * 0= No plaque around the gingival margin.
  * 1= A thin film of plaque around the gingival margin. The plaque may be recognized only by running a probe across the tooth surface.
  * 2= Moderate accumulation of soft deposits on the gingival margin and/or adjacent tooth surface, which can be seen by naked eye.
  * 3= Abundance plaque accumulation within the gingival pocket and/or on the gingival margin and adjacent tooth surface and hard deposits on the tooth surface are seen.
Gingival index (GI) | at base line, 1 month and 3 months after treatment
  It used to assess gingival inflammation. The degree of gingival inflammation was recorded as follow:
  * 0 = Normal gingiva.
  * 1 = Mild inflammation, slight change in color, slight edema and no bleeding on probing.
  * 2= Moderate inflammation, redness, edema and bleeding on probing.
  * 3= Severe inflammation, marked redness, edema and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mortada Fikry, professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao L, Liu G, Wang X, Liu F, Xu Y, Ma J. Preparation of a chemically stable quercetin formulation using nanosuspension technology. Int J Pharm. 2011 Feb 14;404(1-2):231-7. doi: 10.1016/j.ijpharm.2010.11.009. Epub 2010 Nov 17. PMID 21093559
- [Background] Gomez-Florit M, Monjo M, Ramis JM. Quercitrin for periodontal regeneration: effects on human gingival fibroblasts and mesenchymal stem cells. Sci Rep. 2015 Nov 12;5:16593. doi: 10.1038/srep16593. PMID 26558438
- [Background] Wei Y, Fu J, Wu W, Ma P, Ren L, Yi Z, Wu J. Quercetin Prevents Oxidative Stress-Induced Injury of Periodontal Ligament Cells and Alveolar Bone Loss in Periodontitis. Drug Des Devel Ther. 2021 Aug 12;15:3509-3522. doi: 10.2147/DDDT.S315249. eCollection 2021. PMID 34408403
- [Background] Kantarci A, Van Dyke TE. Lipoxin signaling in neutrophils and their role in periodontal disease. Prostaglandins Leukot Essent Fatty Acids. 2005 Sep-Oct;73(3-4):289-99. doi: 10.1016/j.plefa.2005.05.019. PMID 15979867